CLINICAL TRIAL: NCT07117786
Title: Computed Tomography Radiomics-Derived Nomogram for Predicting Early Renal Function Decline After Partial Nephrectomy in Renal Cell Carcinoma: A Multicenter Development/Validation Study
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MRCTA, ECFAH of FMU [2025]570
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: Renal Function Decline; Renal Cell Carcinoma; Computed Tomography
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CT Contrast — Participants will undergo a CT-based radiomics assessment as part of the intervention. This approach involves the extraction of high-dimensional quantitative imaging features from preoperative contrast-enhanced CT scans, which are then analyzed using machine learning algorithms to identify patterns predictive of early postoperative renal function decline. Unlike conventional radiologic evaluations that rely on visual inspection and basic metrics (e.g., tumor size or enhancement), this radiomics-based intervention captures subtle heterogeneity within renal tumors and surrounding parenchyma. The integration of these features with clinical variables distinguishes this study from other imaging or predictive model studies, enabling the development of a personalized nomogram for patients with localized RCC undergoing partial nephrectomy.
Other: Computed Tomography — Participants will undergo a CT-based radiomics assessment as part of the intervention. This approach involves the extraction of high-dimensional quantitative imaging features from preoperative contrast-enhanced CT scans, which are then analyzed using machine learning algorithms to identify patterns predictive of early postoperative renal function decline. Unlike conventional radiologic evaluations that rely on visual inspection and basic metrics (e.g., tumor size or enhancement), this radiomics-based intervention captures subtle heterogeneity within renal tumors and surrounding parenchyma. The integration of these features with clinical variables distinguishes this study from other imaging or predictive model studies, enabling the development of a personalized nomogram for patients with localized RCC undergoing partial nephrectomy.

SUMMARY:
The goal of this observational study is to explore the relationship between CT-based radiomics and postoperative renal function changes in patients with localized renal cell carcinoma (RCC) undergoing partial nephrectomy (PN). The main question it aims to answer is: Can a radiomics-clinical nomogram integrating CT-based radiomics features with preoperative and intraoperative clinical variables accurately predict early postoperative renal function decline in patients with localized RCC undergoing PN? Participants already undergoing renal CT examination and scheduled for postoperative renal function testing as part of the routine perioperative care will receive renal function assessment after completing surgical treatment for RCC.

ELIGIBILITY:
Inclusion Criteria:

* (1) postoperative pathological confirmation of RCC; (2) preoperative contrast-enhanced CT of the kidney or abdomen.

Exclusion Criteria:

* (1) absence of corticomedullary, nephrographic, or excretory phase CT sequences; (2) poor-quality CT images unsuitable for analysis; (3) incomplete clinicopathologic data; (4) missing renal function data during postoperative follow-up; (5) unavailable renal function assessment within two weeks before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was drawn from the following institutions: the First Affiliated Hospital of Fujian Medical University, the Second Affiliated Hospital of Fujian Medical University, the First Affiliated Hospital of Xiamen University, the Second People's Hospital affiliated with Fujian University of Traditional Chinese Medicine, the First Affiliated Hospital of Chongqing Medical University, and Quanzhou First Hospital affiliated with Fujian Medical University
Sampling Method: Probability Sample
Enrollment: 1437 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
early postoperative renal function decline | within 3 to 24 months postoperatively
  early Renal function decline after PN was defined as a ≥25% reduction in eGFR from the preoperative baseline within 3 to 24 months postoperatively

IPD SHARING:
Plan to Share IPD: No